CLINICAL TRIAL: NCT00434447
Title: A Phase IV Study of Zoledronic Acid Therapy in Patients With Bone Metastases From Breast Cancer or Hormone Resistant Prostate Cancer, or Bone Involvement From Multiple Myeloma, Assessing Long-term Efficacy and Safety
Brief Title: Long Term Efficacy and Safety of Zoledronic Acid Treatment in Patients With Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CZOL446EAU22
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2010-10

CONDITIONS: Bone Neoplasms
Keywords: Prostate Cancer; Breast Cancer; Multiple Myeloma; Zoledronic acid; Bone metastases; Skeletal Related Events (SREs); Renal Impairment; Osteonecrosis of the Jaw (ONJ); Bone involvement; Multiple Myeloma (MM)
MeSH Terms: conditions — Bone Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Multiple Myeloma; Renal Insufficiency | interventions — Zoledronic Acid

ARMS (1):
- Zoledronic Acid (Experimental): ZOL446
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
This study is designed to monitor the safety and efficacy of long-term treatment with zoledronic acid by assessing the incidence of, renal impairment, osteonecrosis of the jaw(ONJ), overall safety and skeletal related events (SREs) beyond 12 months treatment

ELIGIBILITY:
Inclusion criteria:

* Documented bone metastases from breast cancer, prostate cancer or multiple myeloma
* Prior treatment with zoledronic acid for 1-2 yrs
* Life expectancy of at least 6 months

Exclusion criteria:

* Prior treatment with bisphosphonates other than zoledronic acid
* Abnormal kidney function
* Current or previous dental problems or planned dental surgery
* Pregnant or likely to become pregnant during the study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of renal impairment, osteonecrosis of the Jaw (ONJ), adverse events and serious adverse events. Efficacy assessed by incidence of skeletal related events (SREs). | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (10):
- Australia (10):
  - Novartis Investigative Site, Canberra, Australian Capital Territory
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Wagga Wagga, New South Wales
  - Novartis Investigative Site, Redcliffe, Queensland
  - Novartis Investigative Site, Townsville, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Ballarat, Victoria
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Frankston, Victoria